CLINICAL TRIAL: NCT06131489
Title: Efficacy and Safety of Segmental Resection Combined With the DEP Regimen for Epstein-Barr Virus Associated Hemophagocytic Lymphohistiocytosis With Intestinal Involvement
Brief Title: Segmental Resection Combined With DEP Regimen for EBV-HLH Patients With Intestinal Involvement
Status: Not yet recruiting | Type: Observational
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Zhao Wang, Professor and Head of hematology, Beijing Friendship Hospital
Other Study IDs: BFH20230809002/BFHHZS20230190
Record Dates: First submitted 2023-11-09; First posted 2023-11-14 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-09

CONDITIONS: Hemophagocytic Lymphohistiocytosis; Epstein-Barr Virus; Bowel Resection
MeSH Terms: conditions — Lymphohistiocytosis, Hemophagocytic; Epstein-Barr Virus Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- EBV-HLH patients with intestinal involvement: Epstein-Barr virus associated hemophagocytic lymphohistiocytosis patients with imaging confirmed intestinal involvement
  Interventions: Other: Segmental bowel resection combined with the DEP regimen

INTERVENTIONS:
Other: Segmental bowel resection combined with the DEP regimen — Segmental bowel resection combined with liposomal doxorubicin, etoposide, and methylprednisolone administered in 2 week cycles for 2 cycles

SUMMARY:
EBV-HLH is a rare disease with high mortality, especially for those with intestinal involvement. In order to reduce disease burden and improve survival of these patients, we conduct a prospective observational study to explore the efficacy and safety of segmental resection combined with the DEP regimen.

DETAILED DESCRIPTION:
Epstein-Barr virus associated hemophagocytic lymphohistiocytosis is a rare disease with high mortality, especially for those with intestinal involvement. Some of them still died despite early control of the disease due to severe complications, such as gastrointestinal bleeding. In order to reduce disease burden and improve survival of these patients, we conduct a prospective observational study to explore the efficacy and safety of segmental resection combined with the DEP regimen.

ELIGIBILITY:
Inclusion Criteria:

* Met HLH-2004 diagnostic criteria;
* EBV-DNA in the peripheral blood > 1000 copies/ml or EBV-encoded small RNA (EBER) detected in tissues;
* Imaging revealed severe intestinal lesions and biopsy confirmed EBV-encoded small RNA (EBER) in the tissues;
* Age >18 years old, gender is not limited;
* Estimated survival time > 1 month;
* Informed consent obtained.

Exclusion Criteria:

* Active infections (viral, bacterial, fungal or parasitic);
* Diagosed with malignant tumos within 5 years；
* Uncontrolled symptoms or other diseases including, but not limited to, unstable angina pectoris, arrhythmia, respiratory failure, severe hepatic or renal insufficiency, severe coagulation dysfunction, mental illness, or other conditions deemed by the attending physician to be contraindications to surgery;
* Heart function above grade II (NYHA);
* Severe myocardial injury：TNT、TNI、CK-MB > 3 ULN;
* Accumulated dose of doxorubicin above 400mg/m2 、epirubicin above 750mg/m2、pirarubicin above 800mg/m2 or the patients treated with anthracycline induced cardiovascular disease;
* Pregnancy or lactating Women;
* Allergic to pegylated liposomal doxorubicin and etoposide;
* HIV antibody positivity;
* Acute or chronic active hepatitis B (HBsAg positivity, HBV DNA negative acceptable), acute or chronic active hepatitis C (HCV antibody negatively acceptable; HCV antibody positivity, HCV RNA negative acceptable);
* Participate in other clinical research at the same time;
* The researchers considered that patients are not suitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: EBV-HLH patients with intestinal involvement
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
ORR | 4 Week
  The percentage of cases that achieved complete response (CR) and partial response (PR) after treatment.
Adverse events | 1 month
  Incidence of adverse reactions

SECONDARY OUTCOMES:
OS | 1 years
  Overall survival rate

CONTACTS AND LOCATIONS:
Overall Officials: Zhao Wang, MD, Principal Investigator — Beijing Friendship Hospital
Locations (1):
- Zhao Wang, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No